CLINICAL TRIAL: NCT02406599
Title: MarginProbe® System U.S. Post-Approval Study Protocol CP-07-001
Brief Title: MarginProbe® System U.S. Post-Approval Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dune Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CP-07-001
Record Dates: First submitted 2015-03-24; First posted 2015-04-02 (Estimated); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOC + Device (Other): The surgeon will perform routine standard of care lumpectomy with adjunctive MarginProbe device use on the main ex-vivo lumpectomy specimen.
  Interventions: Device: Margin Probe
- SOC + Additional Inspection (Other): The surgeon will perform routine standard of care lumpectomy with additional inspection on the main ex-vivo lumpectomy specimen.
  Interventions: Other: Control: Additional inspection

INTERVENTIONS:
Device: Margin Probe — The surgeon will use the MarginProbe System to identify cancerous tissue at the margins (≤ 1mm) of the main ex-vivo lumpectomy specimen following primary excision
  Arms: SOC + Device
Other: Control: Additional inspection — The surgeon will perform additional inspection and assessment of the margins of the main ex-vivo lumpectomy specimen following primary excision
  Arms: SOC + Additional Inspection

SUMMARY:
The study objective is to determine the MarginProbe® System's diagnostic accuracy at the margin level and impact on Positive Margin* Presence originating from the Main ex-vivo lumpectomy specimen after the initial lumpectomy surgery.

*A positive margin is defined in this study as a margin microscopically measured and reported in the histology report to have cancer within 1 mm or less of the inked surface

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized (1:1), double arm, controlled study, in which subjects undergoing breast excision (lumpectomy) for carcinoma of the breast will be randomized to either standard of care with additional inspection ('SOC + Additional inspection' arm) or standard of care with MarginProbe as an adjunct ('SOC + Device' arm).

The MarginProbe is an adjunctive diagnostic tool for identification of cancerous tissue at the margins (≤ 1mm) of the main ex-vivo lumpectomy specimen following primary excision. It will be used by the surgeon during lumpectomy procedures only in patients randomized to the "Device+SOC" arm.

Randomization will take place following the excision of the main ex-vivo lumpectomy specimen.

ELIGIBILITY:
Inclusion Criteria:

* Women histologically diagnosed with carcinoma of the breast
* Women with non-palpable malignant lesions, requiring image guided localization.
* Undergoing lumpectomy (partial mastectomy) procedure
* Age 18 years or more
* Signed ICF

Exclusion Criteria:

* Multi-centric disease (histologically diagnosed cancer in two different quadrants of the breast)
* Bilateral disease (diagnosed cancer in both breasts)
* Neo-adjuvant systemic therapy
* Previous radiation in the operated breast
* Prior surgery in the same site in the breast
* Woman histologically diagnosed by an open biopsy procedure
* Implants in the operated breast
* Pregnancy
* Lactation
* Participating in any other investigational study for either drug or device which could influence collection of valid data under this study
* Patients for whom complete cavity shaving is planned (sites where this is the routine practice of the investigator will also be excluded from participation in the study)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy at the margin level | Participants will be followed only for the initial lumpectomy duration. information will be available 2-3 weeks (avarage) from initial lumpectomy date
  Sensitivity and Specificity at the margin level;
Incomplete Surgical Resection (ISR ) | Participants will be followed only for the initial lumpectomy duration. information will be available 2-3 weeks (avarage) from initial lumpectomy date
  ISR - Positive Margin on the Main ex-vivo lumpectomy specimen after the initial lumpectomy surgery, that was not addressed by taking a shaving(s) corresponding to the positive margin(s).

SECONDARY OUTCOMES:
Positive Margin presence on the Outermost Shaving after the initial lumpectomy surgery | Participants will be followed only for the initial lumpectomy duration. information will be available 2-3 weeks (avarage) from initial lumpectomy date
  Proportion of patients with Positive Margin presence on the Outermost Shaving after the initial lumpectomy surgery
Cosmesis evaluation | participants will be followed until 6 months ± 1 month after last surgical treatment visit, an avarage of of 8 months following initial lumpectomy
  Objective evaluation by an evaluator blinded to arm assignment
Repeat lumpectomy rate | Participants will be followed for 2-5 weeks (average)
  Proportion of patients who underwent a repeat lumpectomy procedure
Repeat lumpectomy and mastectomy rate | Participants will be followed for 2-5 weeks (average)
  Proportion of patients who underwent a repeat lumpectomy procedure or a mastectomy
Diagnostic Accuracy at the Patient Level (ignoring location) | Participants will be followed only for the initial lumpectomy duration. information will be available 2-3 weeks (avarage) from initial lumpectomy date
  Proportion of patients from whom shavings were taken

CONTACTS AND LOCATIONS:
Overall Officials: Maya Livnat, Study Director — Dilon Medical Technologies Ltd.
Locations (11):
- United States (11):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - NorthShore University HealthSystem, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - John Hopkins Medicine, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Summit Medical Group, Berkeley Heights, New Jersey
  - New Mexico University Cancer center, Albuquerque, New Mexico
  - Montefiore Medical Center, New York, New York
  - PinnacleHealth Cancer Institute, Harrisburg, Pennsylvania

REFERENCES:
- See also: A randomized prospective study of lumpectomy margin assessment with use of MarginProbe in patients with nonpalpable breast malignancies. — http://www.ncbi.nlm.nih.gov/pubmed/24595800
- See also: Dune Medical Devices official website — http://www.dunemedical.com